CLINICAL TRIAL: NCT00004306
Title: Pathogenic Mechanism of Spinocerebellar Ataxia Type 10 (SCA10)
Brief Title: Clinical and Molecular Correlations in Spinocerebellar Ataxia Type 10 (SCA10)
Status: Completed | Type: Observational
Sponsor: Office of Rare Diseases (ORD) (NIH)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Principal Investigator, Tetsuo Ashizawa, Professor and Chair, Department of Neurology, The University of Texas Medical Branch, Office of Rare Diseases (ORD)
Other Study IDs: 199/11796
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Hereditary Ataxia
Keywords: hereditary ataxia; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Spinocerebellar Degenerations; Neurologic Manifestations; Mental Disorders; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood and skin and muscle biopsy samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
OBJECTIVES: I. Clinically evaluate members from families with a dominantly inherited ataxia and collect blood, skin and muscle samples for detailed molecular studies.

II. Perform detailed clinical evaluations on patients with recessively inherited ataxias.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants undergo a comprehensive clinical and molecular evaluation. Studies include: neurologic evaluation, including magnetic resonance imaging and nerve conduction studies; ophthalmologic exam; audiologic exam, including auditory brain stem evoked response; DNA extraction from blood, skin and muscle; genotype phenotype correlation.

A neuropathologic evaluation is conducted postmortem, when possible.

ELIGIBILITY:
Inclusion criteria:

Subjects who have the diagnosis of SCA10 and their immediate relatives.

Exclusion criteria:

Children under 3 years of age, pregnant women, prisoners, mentally incapacitated subjects, and subjects who do not give consent.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inherited ataxia
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 1999-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuo Ashizawa, MD, Principal Investigator — University of Texas, Galveston
Locations (1):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States